CLINICAL TRIAL: NCT04295486
Title: Optimal Dosing For Low-Dose Aspirin Chemoprophylaxis For Venous Thromboembolism (VTE) Following Total Joint Arthroplasty - A Multi-center Prospective Randomized Control Trial.
Brief Title: Optimal Dosing For Low-Dose Aspirin Chemoprophylaxis For VTE Following Total Joint Arthroplasty
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Victor Hugo Hernandez, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20190973
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Venous Thromboembolism
Keywords: Chemoprophylaxis; Hip Surgery; Knee Surgery
MeSH Terms: conditions — Venous Thromboembolism | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Once Daily (Experimental): Participant receives 81 mg aspirin taken once daily beginning the night before surgery and up to 28 days post surgery.
  Interventions: Drug: Aspirin
- Treatment Twice Daily (Active Comparator): Participant receives 81 mg aspirin taken twice daily (one in the morning and one at night) beginning at the night before surgery and up to 28 days post surgery.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Non-enteric coated 81 mg Aspirin tablet.

SUMMARY:
This research study is attempting to answer the question of whether 81 mg aspirin once daily is as effective as 81 mg aspirin twice daily in preventing blood clots after total joint replacement surgery.

ELIGIBILITY:
Inclusion criteria:

* > 18 years of age
* Planning to undergo a primary total hip or knee arthroplasty

Exclusion Criteria:

* High risk patients for VTE as defined by:

  * History of venous thromboembolism
  * Active malignancy
  * Known pro thrombotic condition
* BMI > 40
* Patients requiring anticoagulation for pre-existing conditions
* Patients with the contraindication for use of aspirin or nonsteroidal antiinflammatory drugs for reasons such as peptic ulcer disease, intolerance, others.
* Patients not fluent in the language of the informed consent form
* Prisoners
* Pregnancy
* Reported to have mental illness or belonging to a vulnerable population

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5478 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of symptomatic thromboembolic events | 90 days
  Efficacy of prophylaxis will be reported as the number of reported incidence of symptomatic Pulmonary Embolism (PE) and Deep Vein Thrombosis (DVT).

SECONDARY OUTCOMES:
Incidence of specific adverse events | 90 days
  Efficacy of prophylaxis will be reported as the number of reported incidence of specific adverse events including gastrointestinal (GI) complications, post-operative hematoma, bleeding and wound complications and infections.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Hernandez, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No